CLINICAL TRIAL: NCT07114653
Title: The Role of POLE Mutation in High Risk Endometrial Cancer.
Status: Recruiting | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 113298-E
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Endometrial Neoplasms
Keywords: Endometrial cancer; POLE mutation
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- endometrial cancer: high-risk for reurrence of endometrial cancer.

SUMMARY:
The actual role of POLE mutations in high-risk endometrial cancer is undetermined. The main question it aims to answer is:

What is the prevalence of POLE mutations in high-risk endometrial cancer case? What is the impact of POLE mutations in real world high-risk endometrial cancer case?

DETAILED DESCRIPTION:
All high-risk recurrent endometrial cancer cases who were treated in a tertiary referral center will be analyzed and subjected to POLE mutation analysis. In addition, survival analysis will be used to analyze the role of POLE mutations in women with high-risk endometrial cancer. We can answers the following.

1. What is the prevalence of POLE mutations in women with high-risk endometrial cancer?
2. What is the role of POLE mutations in real world high-risk endometrial cancer?

ELIGIBILITY:
Inclusion Criteria:

* women with high-risk for recurrent endometrial cancer

Exclusion Criteria:

* Nil

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — women with high-risk endometrial cancer
Study Population: All high-risk endometrial cancer cases
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of POLE mutation in high risk endometrial cancer | 2 years
  The prevalence of POLE mutations in women with high-risk for recurrent endometrial cancer

SECONDARY OUTCOMES:
The impact of POLE on overall survival | 5 years
  The impact of POLE on overall survival, compared with the other TCGA groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No